CLINICAL TRIAL: NCT00692367
Title: Physical Activity Following Surgery Induced Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: East Carolina University (Other)
Responsible Party: Principal Investigator, Bret Goodpaster, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO007090041; R01DK078192-01A1 (NIH)
Record Dates: First submitted 2008-06-02; First posted 2008-06-06 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Obesity
Keywords: Body fat; Exercise; Fatty acids; Impaired glucose tolerance; Insulin resistance; Insulin Sensitivity; Metabolic syndrome; Obesity; Physical activity; Weight Loss
MeSH Terms: conditions — Obesity; Motor Activity; Glucose Intolerance; Insulin Resistance; Metabolic Syndrome; Weight Loss | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exercise (Other): Structured exercise program
  Interventions: Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Physical Activity — 1. Physical activity group: Subjects will be progressed to 4-5 days per week, 30-45 min per session (120-180 min per week) of moderate intensity exercise. 2. Control (educational) group: Subjects will receive their usual care following surgery that in addition to their weight loss.

SUMMARY:
The primary objective of this study will be to determine the effects of physical activity in patients during substantial surgery-induced weight loss.

A randomized controlled physical activity intervention trial in a group of patients undergoing bariatric surgery for weight loss. The study will involve two sites with an active bariatric surgery program, which have a strong track record of bariatric surgery research. The study will include 160-200 subjects. Changes in the primary outcome variables will be determined in previous gastric bypass patients as a result of 6 months of moderate physical activity compared to an educational control group not engaged structured exercise.

DETAILED DESCRIPTION:
The primary objective of this study will be to determine the effects of physical activity in patients during substantial surgery-induced weight loss. We propose to employ a randomized controlled physical activity intervention trial in a group of patients undergoing bariatric surgery for weight loss. The study will involve two sites with an active bariatric surgery program, which have a strong track record of bariatric surgery research.

Recruitment goals are 160-200 gastric bypass patients who will undergo 6 months of moderate physical activity compared to an educational control group not engaged structured exercise. Subjects will be included if their BMI is less than 55 kg/m2 prior to surgery and they are located relatively close to centers for intervention sessions. At baseline (3 months following surgery) and 6 months later (9 months following surgery), subjects will have a CT scan, IV glucose tolerance test (IVGTT) and muscle biopsy (~8 hour visit). They will be scheduled for separate visits for a test of physical fitness (VO2max) and general body composition (DXA scan)(~2 hour visit), and a 15-min sub-maximal exercise session.

1. Physical activity group: Subjects will be progressed to 4-5 days per week, 30-45 min per session (120-180 min per week) of moderate intensity exercise.
2. Control (educational) group: Subjects will receive their usual care following surgery that includes information on physical activity. They will also be asked to participate in monthly health education sessions.

We will promote this study as one that will help determine whether physical activity may be beneficial in addition to their weight loss.

Aim 1: Insulin resistance and metabolic risk factors. Approach: To address Aim 1, we will determine 6-month changes in insulin sensitivity in subjects after 3-month initial weight loss from bariatric surgery. As outlined above, we will employ a randomized controlled physical activity intervention trial in which half of the subjects will be entered into a physical activity group, while the other half will participate in monthly health education sessions (control). By randomizing these groups three months after initial weight loss, both groups should begin the intervention with similar baseline characteristics (e.g. insulin sensitivity, body weight, physical fitness, etc.). We are not attempting to determine the effect of the weight loss per se on insulin sensitivity. However, we realize that the amount of weight loss could potentially have a major confounding influence on detecting changes in insulin sensitivity between the two groups. Thus, we will examine the degree of weight loss as a covariate in our analyses.

Aim 2: Intramyocellular lipids and body composition. Approach: We will examine pre to post intervention, changes in intramyocellular lipid determined with percutaneous biopsies, as well as abdominal and intermuscular adipose tissue determined by CT imaging.

Aim 3: Mitochondria content, function and fat oxidation. Approach: We will use three complimentary measures to quantify changes in oxidative metabolism before and after the randomized controlled trial described above. All three of these measures will make specific contributions to this specific aim. Rates of resting post-absorptive fat oxidation will be measured with indirect calorimetry. Since skeletal muscle accounts for the vast majority of energy production during physical activity, sub-maximal exercise is a good model to assess skeletal muscle fatty acid metabolism. We will employ whole body gas exchange indirect calorimetry during moderate exercise designed to elicit high rates of fatty acid oxidation. The non-invasive measures of systemic fat oxidation during both resting and exercise conditions procedures take very little time and present relatively little burden on the volunteers or technical staff, thus providing an efficient means to obtain significant information concerning the capacity for fat oxidation in vivo. Muscle biopsy samples will be obtained before and after the trial to measure changes in the oxidative capacity (electron transport chain activity, in vitro fatty acid oxidation, muscle fiber type and oxidative enzyme (succinate dehydrogenase) staining activity of muscle.

ELIGIBILITY:
Inclusion Criteria:

* Men and women (21-60 years of age) good health, stable weight, and without any contraindication to exercise.

Exclusion Criteria:

* Anemia (Hct<34%)
* Elevated liver enzyme (25% above normal),
* Proteinuria,
* Hypothyroidism (sTSH > 8)
* Hypertension (blood pressure > 150 mmHg systolic, or > 95 mmHg diastolic)
* Diabetes mellitus (fasting glucose ≥ 126 mg/dl)
* A history of myocardial infarction or peripheral vascular disease
* Liver disease
* Alcohol or drug abuse
* Malignancy or neuromuscular disease
* Subjects will be excluded if taking chronic medications known to adversely affect glucose homeostasis (oral glucocorticoids, nicotinic acid)
* Females currently on hormone replacement therapy (HRT) can participate in the study if they have been on HRT for at least 6 months and will continue to be on HRT during the study.
* Disqualifying findings on physical examination include:

  * Lower extremity thrombophlebitis
  * Evidence of peripheral neuropathy, paresis or edema.

If the resting EKG prior to the exercise test shows any abnormalities, the test will not be conducted. If any abnormalities develop during the test, the test will be stopped. On both occasions, the participant will be referred to their PCP for further evaluation and will only be allowed to continue the study with written clearance by his/her PCP or cardiologist. American College of Sports Medicine (ACSM) criteria will be used to halt maximal exercise testing should adverse cardiovascular responses develop. Only after a cardiologist interprets the resting and exercise ECG of the participant and clears them for exercise, will subjects be able to continue with the study

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2007-12; Primary Completion 2011-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity, intramyocellular lipid, total body fat, total lean mass | Twelve months

SECONDARY OUTCOMES:
Intra-muscular adipose tissue, abdominal fat, mitochondria content, fat oxidation | Twelve months

CONTACTS AND LOCATIONS:
Overall Officials: Bret H Goodpaster, Ph.D., Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - East Carolina University, Greenville, North Carolina
  - Montefiore Hospital, N807, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Carnero EA, Dubis GS, Hames KC, Jakicic JM, Houmard JA, Coen PM, Goodpaster BH. Randomized trial reveals that physical activity and energy expenditure are associated with weight and body composition after RYGB. Obesity (Silver Spring). 2017 Jul;25(7):1206-1216. doi: 10.1002/oby.21864. Epub 2017 May 30. PMID 28558160
- [Derived] Nunez Lopez YO, Coen PM, Goodpaster BH, Seyhan AA. Gastric bypass surgery with exercise alters plasma microRNAs that predict improvements in cardiometabolic risk. Int J Obes (Lond). 2017 Jul;41(7):1121-1130. doi: 10.1038/ijo.2017.84. Epub 2017 Mar 27. PMID 28344345
- [Derived] Coen PM, Menshikova EV, Distefano G, Zheng D, Tanner CJ, Standley RA, Helbling NL, Dubis GS, Ritov VB, Xie H, Desimone ME, Smith SR, Stefanovic-Racic M, Toledo FG, Houmard JA, Goodpaster BH. Exercise and Weight Loss Improve Muscle Mitochondrial Respiration, Lipid Partitioning, and Insulin Sensitivity After Gastric Bypass Surgery. Diabetes. 2015 Nov;64(11):3737-50. doi: 10.2337/db15-0809. Epub 2015 Aug 20. PMID 26293505
- [Derived] Coen PM, Tanner CJ, Helbling NL, Dubis GS, Hames KC, Xie H, Eid GM, Stefanovic-Racic M, Toledo FG, Jakicic JM, Houmard JA, Goodpaster BH. Clinical trial demonstrates exercise following bariatric surgery improves insulin sensitivity. J Clin Invest. 2015 Jan;125(1):248-57. doi: 10.1172/JCI78016. Epub 2014 Dec 1. PMID 25437877